CLINICAL TRIAL: NCT00836134
Title: Ultrasound-guided Rectus Sheath Block for Post-operative Pain Control Following Umbilical Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Sean Flack, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RS_Rectus_sheath
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2014-06-12 (Estimated); Status verified 2014-06

CONDITIONS: Pain
Keywords: pain relief after umbilical hernia repair; morphine consumption; plasma bupivacaine levels
MeSH Terms: conditions — Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): rectus sheath block
  Interventions: Procedure: rectus sheath block
- 2 (Active Comparator): local anesthetic infiltration
  Interventions: Procedure: local anesthetic infiltration

INTERVENTIONS:
Procedure: rectus sheath block — ultrasound-guided rectus sheath block using 0.2ml/kg 0.25% bupivacaine bilaterally prior to skin incision
  Other Names: bupivacaine
  Arms: 1
Procedure: local anesthetic infiltration — Wound infiltration using 0.4ml/kg 0.25% bupivacaine by the surgeon at the end of surgery
  Other Names: bupivacaine
  Arms: 2

SUMMARY:
The purpose of this study is to compare the effectiveness of local infiltration to an ultrasound guided nerve block placed by the anesthesiologist for children undergoing umbilical hernia repair.

This is a double-cohort, double blinded, randomized study comparing local infiltration to ultrasound-guided rectus sheath block in children 1 to 17 years of age undergoing epigastric or umbilical hernia repair.

We will first compare pain scores to see if one method is more adequate then the other in providing post-op analgesia. Our second aim is to compare morphine consumption between the two groups.

Our third aim is to measure the levels of local anesthetic in the blood following local anesthetic infiltration or USGRSB.

DETAILED DESCRIPTION:
Healthy children, aged 1 to 17 years of age, undergoing elective umbilical hernia repairs will be considered for this study. After informed consent/assent has been obtained, the subject will be randomized into one of two groups. Group A will receive local infiltration of 0.25% bupivacaine by the surgeon at the end of the subject's surgery. Group B will undergo an ultrasound-guided rectus sheath block using 0.25% bupivacaine prior to incision by an anesthesiologist skilled in the performance of this block.

All subjects will receive a standardized anesthetic for their surgery. Subjects assigned to Group A (local infiltration) will receive 2mcg/kg of fentanyl prior to incision for intra-operative pain management. Subjects assigned to Group B will have their Rectus Sheath Block and no fentanyl will be given at this time.

Fentanyl is a short-acting opioid analgesic. It's duration of action in the dose we will be using is approximately one hour which is close to the expected length of surgery. Therefore, it is not expected to influence the pain management after surgery.

Pain scores will be assessed by a member of the research team. They will be blinded to which technique the subject has been randomized to. This person will not be involved in the direct care of the subject. These observations will be made using an age-appropriate scoring system (FLACC or FACES scale). Scoring will be done every 5 minutes when the subject is in the recovery room and every 30 minutes when they are in Phase II. This will be done until the subject is discharged from the hospital.

Families will be followed by phone for 48 h post discharge, to collect data on medication use.

ELIGIBILITY:
Inclusion Criteria:

* Children between 1 ≤ 17 years of age
* ASA I (normal healthy children) and II (Children with mild systemic disease that has no functional effects)
* Having elective umbilical hernia repair

Exclusion Criteria:

* Children < 1 year of age or > 17 years of age
* Family has no telephone for follow up phone call
* Allergy or sensitivity to bupivacaine or morphine
* Any coagulation abnormalities
* Emergency surgery

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
pain scores | 4 hours

SECONDARY OUTCOMES:
morphine consumption | 4 hours
plasma bupivacaine levels | 0, 10, 20, 30, 45, 60 minutes after injection

CONTACTS AND LOCATIONS:
Overall Officials: Sean H Flack, MBChB FCA, Principal Investigator — University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States